CLINICAL TRIAL: NCT01748812
Title: Open-label Dose-titration Study of the Tolerability and Efficacy of Cinacalcet to Treat Fibroblast Growth Factor 23 (FGF23)-Mediated Hypophosphatemia
Brief Title: Cinacalcet for Fibroblast Growth Factor 23 (FGF23)-Mediated Hypophosphatemia (Hypophosphatemic Rickets)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 130025; 13-D-0025
Record Dates: First submitted 2012-12-11; First posted 2012-12-13 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2015-07-07

CONDITIONS: Osteomalacia
Keywords: Tumor Induced Osteomalacia; Hypophosphatemic Rickets
MeSH Terms: conditions — Osteomalacia; Oncogenic osteomalacia; Rickets, Hypophosphatemic

INTERVENTIONS:
Drug: Osteomalacia

SUMMARY:
Background:

* Hypophosphatemia is a condition where a person has low levels of phosphorus in the blood. Low blood phosphorus can cause muscle and bone weakness (such as rickets) and teeth problems. One cause of the condition is having too much fibroblast growth factor 23 (FGF23). FGF23 is a hormone that causes the kidney to get rid of phosphorus in the urine. It can also prevent the body from making vitamin D, which helps the body absorb phosphorus in food.
* Many people with low blood phosphorus take high doses of phosphorus and calcium medications. However, one side effect of these drugs is increased blood levels of parathyroid hormone (PTH). The drug cinacalcet can help lower PTH levels, which may decrease the amount of phosphorus lost in the urine and increase the phosphorus levels in the blood. Researchers want to see if cinacalcet can help blood phosphorus and decrease the amount of phosphorus supplements that people need to take.

Objectives:

- To see if cinacalcet can be a safe and effective treatment for people with low phosphorus conditions due to high FGF23.

Eligibility:

- Individuals between 18 and 70 years of age who have different forms of hypophosphatemic rickets and tumor-induced hypophosphatemia

Design:

* Participants will have up to 25 study visits over about 28 weeks.
* Participants will be screened with a physical exam and medical history. Blood and urine samples will be collected.
* Up to three more lab visits for blood and urine tests will be required before treatment. Imaging studies of the bones, spine, and kidneys will be performed.
* Participants will have a 3-night hospital stay to start treatment. They will take cinacalcet once a day. Treatment will be monitored with frequent blood tests and imaging studies.
* Participants will continue to take cinacalcet once a day for 3 weeks. They will have regular study visits to monitor the treatment.
* There will be up to two other overnight hospital stays (1 to 3 nights) to adjust cinacalcet doses. The dose will increase until the maximum dose is reached, or side effects develop.
* After the end of the cinacalcet study, participants will have several more followup visits to monitor the effects of treatment.

DETAILED DESCRIPTION:
OBJECTIVES:

The primary objective of this protocol is to evaluate the tolerability of cinacalcet in individuals with fibroblast growth factor 23 (FGF23)-mediated hypophosphatemia, using an open-label, dose-titration study of once-daily dosing. Secondary objectives are to evaluate the pharmacodynamics of cinacalcet in this subject population and to explore the efficacy of cinacalcet by comparing a) level of oral phosphate required at baseline to the level required at maximum tolerated dose (MTD) and b) change in renal phosphate handling from baseline to MTD. Tertiary objectives are to evaluate tolerability, pharmacodynamics, and efficacy of twice daily dosing of each subject s MTD of cinacalcet after completion of the once-daily dose-titration phase. A final objective is to determine the length of time it takes for subjects to return to their pre-treatment steady state once treatment is complete.

STUDY POPULATION:

Up to 17 subjects with FGF23-mediated hypophosphatemia will be treated.

DESIGN:

This study is an open-label, dose-titration study of once-daily dosing of cinacalcet, with up to 4 escalating doses given at approximately 3 week intervals. After an initial standard of care optimization period of 2-9 weeks, subjects will proceed to the cinacalcet dose-titration period. Subjects who experience extended toxicity or study drug related serious adverse events or other related, intolerable adverse events will be down titrated to a lower dose of study medication. After subjects have achieved their own maximum tolerated dose (MTD) and completed the once-daily dosing phase, they will continue the study medication for approximately 3 additional weeks with twice daily dosing at their MTD. At the end of the cinacalcet treatment phase of the study, cinacalcet will be discontinued and standard of care (SOC) medications will be adjusted/restarted on an individualized basis. Subjects will continue in this final SOC safety follow-up period for up to 4 weeks until their SOC medications have been re-equilibrated.

OUTCOME MEASURES:

Primary safety:

Whether or not a subject discontinued the study due to a toxicity, related serious adverse event (SAE), or related intolerable adverse event (AE).

Secondary safety:

* <TAB>Maximum tolerated dose of cinacalcet
* <TAB>Serum calcium levels
* <TAB>Urine calcium levels
* <TAB>Adverse events
* <TAB>Time from cinacalcet discontinuation to return to pre-treatment standard of care dosage levels

Secondary efficacy:

* <TAB>Pharmacodynamic assessments
* <TAB>Serum: FGF23, intact parathyroid hormone, calcium, creatinine, phosphorus
* <TAB>Urine: phosphorus, creatinine, calcium.
* <TAB>Tubular maximum reabsorption of phosphate/glomerular filtration rate
* <TAB>Tubular reabsorption of phosphate
* <TAB>Other
* <TAB>Change in oral phosphate and calcitriol intake required to maintain adequate phosphorus and calcium serum levels
* <TAB>Serum osteocalcin and alkaline phosphatase
* <TAB>Serum intact parathyroid hormone (PTH)

Tertiary efficacy:

* <TAB>Twice-Daily Dosing at MTD
* <TAB>Time from cinacalcet discontinuation of twice-daily dosing to return to pre-treatment standard of care dosage levels
* <TAB>Dental Evaluation
* <TAB>Visible Plaque Index (VPI)
* <TAB>Gingival Bleeding Index (GBI)
* <TAB>Position of Gingival Margin (PGM)
* <TAB>Relative Attachment Level (RAL)
* <TAB>Periodontal Probing Pocket Depth (PPD)
* <TAB>Gingival Crevicular Fluid (GCF) Biomarkers

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. <TAB>Chronological age: 18-70 years
  2. <TAB>Diagnosis of a genetic form of FGF23-mediated hypophosphatemia:

     1. <TAB>X-linked hypophosphatemic rickets (XLH)
     2. <TAB>Autosomal dominant hypophosphatemic rickets (ADHR)
     3. <TAB>Autosomal recessive hypophosphatemic rickets (ARHR)

     Or, diagnosis of a non-genetic form of FGF23-mediated hypophosphatemia, i.e. tumor-induced osteomalacia (TIO)
  3. <TAB>Ability to understand and provide informed consent
  4. <TAB>Ability to complete the protocol scheduled assessments and medication regimen
  5. <TAB>Women of child-bearing potential (not surgically sterile via tubal ligation, bilateral oophorectomy or hysterectomy, or who are not postmenopausal for greater than or equal to 1 year) must agree to practice adequate contraception that may include, but is not limited to, abstinence, monogamous relationship with vasectomized partner, barrier methods such as condoms, diaphragms, spermicides, intrauterine devices, and licensed hormonal methods for the duration of the treatment portion of the study.

EXCLUSION CRITERIA:

1. <TAB>Chronic or recurrent hypocalcemia defined by a serum calcium < 8.4 mg/dL (2.1 mmol/L)
2. <TAB>Tertiary hyperparathyroidism as evidenced by concurrent PTH and calcium levels above the upper limit of normal
3. <TAB>History of parathyroid surgery and/or hypoparathyroidism
4. <TAB>Hypercalciuria as defined as > 4 mg/kg/day (0.1 mmol/kg/day) on optimized conventional therapy (as determined during SOC optimization phase)
5. <TAB>Moderate to severe hepatic insufficiency as defined by total bilirubin > 2 mg/dL and serum albumin < 3 g/dL and International Normalized Ratio (INR) >2 OR presence of ascites or hepatic encephalopathy.
6. <TAB>A calculated eGFR < 50 mL/min/1.73 m(2), using the CKD-EPI equation
7. <TAB>History of a non-febrile seizure disorder
8. <TAB>History of a clinically significant cardiac arrhythmia
9. <TAB>History of chronic gastrointestinal disease
10. <TAB>Current therapy (at the time of informed consent) bisphosphonates, calcitonin, diuretics or medications that may have a significant drug interaction with cinacalcet
11. <TAB>Known hypersensitivity to cinacalcet or any of its constituents
12. <TAB>Positive pregnancy test or lactation
13. <TAB>Use of another investigational agent (i.e., in the context of a clinical trial, use of an investigational product that may have impact on the study) within the last 3 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2012-11-16; Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Evaluate the tolerability of cinacalcet in individuals with FGF23-mediated hypophosphatemia | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Rachel I Gafni, M.D., Principal Investigator — National Institute of Dental and Craniofacial Research (NIDCR)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Chen L, Liu H, Sun W, Bai X, Karaplis AC, Goltzman D, Miao D. Fibroblast growth factor 23 overexpression impacts negatively on dentin mineralization and dentinogenesis in mice. Clin Exp Pharmacol Physiol. 2011 Jun;38(6):395-402. doi: 10.1111/j.1440-1681.2011.05526.x. PMID 21488937
- [Background] Makitie O, Doria A, Kooh SW, Cole WG, Daneman A, Sochett E. Early treatment improves growth and biochemical and radiographic outcome in X-linked hypophosphatemic rickets. J Clin Endocrinol Metab. 2003 Aug;88(8):3591-7. doi: 10.1210/jc.2003-030036. PMID 12915641
- [Background] Bastepe M, Juppner H. Inherited hypophosphatemic disorders in children and the evolving mechanisms of phosphate regulation. Rev Endocr Metab Disord. 2008 Jun;9(2):171-80. doi: 10.1007/s11154-008-9075-3. Epub 2008 Mar 26. PMID 18365315